CLINICAL TRIAL: NCT06674161
Title: The Impact of Type 2 Diabetes Mellitus on Cardiovascular Events in Saudi Arabia Now and Future
Status: Not yet recruiting | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Fahad Ahmed Wali, Consultant, Endocrinology, King Faisal Specialist Hospital & Research Center
Other Study IDs: RAC/M 2024-31
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Mortality of Patients with CVD; Mortality of Patients with CVD and T2DM; Mortality of Patients with T2DM; Mortality of Patients with Neither; Morbidity of CVD; Cardiovascular Diseases; Cardiovascular Diseases Risk
Keywords: CVD; T2DM; mortality; morbidity; CVD risk
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- CVD with type 2 diabetes
- CVD without type 2 diabetes
- T2DM only without CVD
- No T2DM and no CVD

SUMMARY:
Cardiovascular disease (CVD) and Type 2 diabetes mellitus (T2DM) are major global health challenges with significant morbidity and mortality. In Saudi Arabia, the prevalence of CVD and T2DM is increasing. This poses a significant burden on the healthcare system. Despite extensive global research, there remains a lack of comprehensive studies examining the combined impact of CVD and T2DM in the Saudi population, particularly in the Western region. Objectives: The primary objectives of the study are: (1) quantify the incidence and mortality rates of CVD and T2DM across various demographics in the Western region of Saudi Arabia; (2) analyse the demographic, clinical, and lifestyle factors contributing to cardiovascular risk in individuals with both conditions; (3) understand the influence of cultural, social, and religious beliefs on health behaviours related to CVD and T2DM using social media and survey data; (4) develop a predictive model for forecasting future cardiovascular events in the Saudi population; and (5) evaluate the impact of the ICD11 classification of CVD. Methodology: The project will include team of experts from King Faisal Specialist Hospital and Research Centre, Madinah, Taibah University, Islamic University of Madinah, University of Prince Mugrin, and King's College University, London. We will work under four workstreams (WS) which are: WS 1: This group will supervise the data collection, analysis and ensure efficient running of the project. WS 2: In year 1, retrospective data will be collected on the service needs, long term outcomes, and mortality of patients with CVD and T2DM, CVD only, T2DM only, and neither. Between Year 1 to 5, we will collect data prospectively using the new ICD-11 criteria. Both, retrospective and prospective data will be used to develop an artificial intelligence (AI) based predictive model. WS 3: Social media survey will be undertaken to understand health beliefs and behaviours influencing health related outcome to CVD and T2DM. WS 4: Undertake economic analyses into long-term resource utilisation and cost of care for CVD and T2DM.

Expected Outcomes:

The study is expected to provide a detailed incidence and all-cause mortality CVD and T2DM in the Western region of Saudi Arabia. This will help in identifying risk factors and predictive for CVD and understand health beliefs and behaviours in Saudi Arabia. The data will help in developing policies, guidelines and awareness programmes in collaboration with policy makers. In conclusion, this study will impact by improving epidemiological knowledge and understanding of CVD and T2DM in Saudi Arabia. The project will support the overall mission of Saudi Vision 2030 with regard to increasing the health and well-being of the population.

DETAILED DESCRIPTION:
Innoviation:

The proposed study will introduce a novel theoretical framework and methodology for comprehensive investigation of the interrelationship between the various combinations of CVD and T2DM within Saudi Arabia.

Key features of the innovative theoretical concept include:

1. Population specific focus: Our research will be focused on the population of Saudi Arabia based demographic, cultural and environmental factors influencing the incidence and outcomes of CVD and T2DM.
2. Health belief: Our study will investigate health beliefs and behaviour related to CVD and T2DM. This would involve using artificial intelligence data analytic per direct questionnaires, published literature, and social media.
3. Predictive modelling: We aim to conduct a predictive modelling and develop a functional model that predicts future CVE and diabetes related cardiovascular complications.

Key innovative methodologies and approaches include:

1. Retrospective population-based study: A large population-based retrospective study will be conducted to determine the incidence and mortality of CVD with and without T2DM. This methodology will thus provide robust epidemiological data by adjusting for possible confounders using Cox regression models in determining hazard ratios.
2. Combination of CVD with/without T2DM: The results will be compared across the four groups: individuals with no CVD and T2DM, CVD only, T2DM only, and both conditions.
3. Risk factor insight: Understanding the risk factors concerning CVD and T2DM in Saudi Arabia.
4. Using AI to evaluate health belief: Conducting large scale survey on health belief using AI to analyse data obtained from existing literature, digital resources, social media platforms, and direct questionnaires.
5. Development of predictive model for future CV events: This model will be based on detailed analysis and interpretation of collected data. This will facilitate the forecasting of disease patterns and guiding preventive approaches.
6. Collaborative approach: The project involves a collaborative effort by experts from King Faisal Specialist Hospital and Research Centre, Madinah, Taibah University, Islamic University of Madinah, University of Prince Mugrin, and King's College University, London. This multidisciplinary approach ensures a comprehensive analysis that utilises diverse expertise

Methodology:

Aims and objectives We aim to improve the lives of people with CVD, T2DM and other risk factors through innovative data collection, use of data, and design personalised and optimised management strategies. We will accomplish this by creating four workstreams (WS), which will run in parallel and work collaboratively throughout the programme.

1. Workstream 1 (WS1): We will engage with those who have suffered from CVD. They will grouped into three main groups: those with Stroke, IHD and other CVD. The three groups will be subdivided into two subcategories: those with and without T2DM. This group will have individuals who are survivors of this disease, carers, public health experts, clinicians and policymakers. This group will shape the data collection, analysis and use of the data.
2. Workstream 2 (WS2): We will work towards estimating the impact of the WHO ICD11 definition of stroke, atherosclerotic CAD and T2DM. The group will also try to understand the long-term outcome and care needs of CVD survivors both individually and as a population.
3. Workstream 3 (WS3): We will use social media, community forums and healthcare facilities to understand the health beliefs of the individual and population groups. We will try to understand the effect on the health outcome of the individual and the population of these health beliefs.
4. Workstream 4 (WS4): This stream will estimate the economic impact of care, service models, and options with the aim of improving decision-making for policymakers, survivors, and individuals at higher risk, as well as their families.

ELIGIBILITY:
Inclusion Criteria:

All adult patients with available records in the western region of Saudi Arabia

Exclusion Criteria:

age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients in the western region of Saudi Arabia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study | 12 months
  Quantify the incidence, trends, and mortality rates of CVD and T2DM across different regions and demographics in the western region of Saudi Arabia,

SECONDARY OUTCOMES:
Risk Factors Evaluation | 24 months
  * Analyse various demographic, clinical, and lifestyle factors contributing to cardiovascular risk in individuals with CVD and T2DM to indicate inequalities among different phenotypes and identify critical risk factors for targeted prevention and management.
  * Understand cultural, social, and religious factors that influence health beliefs and perceptions related to CVD and T2DM using data from social media in Saudi Arabia. This will facilitate the design of culturally appropriate health interventions.

OTHER OUTCOMES:
Predictive Model | 36 Months
  Develop a predictive model to forecast future CVD events across various combinations of CVD and T2DM. This will provide early individualized management to improve secondary prevention. The data from this modelling work will provide key insights to support self-management via an already existing electronic patient portal.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Al-Jedai A, Almudaiheem H, Al-Salamah T, Aldosari M, Almutairi AR, Almogbel Y, AlRuthia Y, Althemery AU, Alluhidan M, Roudijk B, Purba FD, Awad N, O'jeil R. Valuation of EQ-5D-5L in the Kingdom of Saudi Arabia: A National Representative Study. Value Health. 2024 May;27(5):552-561. doi: 10.1016/j.jval.2024.01.017. Epub 2024 Feb 9. PMID 38342365
- [Background] Jatoi NA, Elamin YA, Said AH, Al-Namer B, Al-Muallim FA, Al-Nemer FF, Al-Halal FM. Prevalence of Cardiovascular Risk Factors Among Patients With Diabetes Mellitus Type 2 at King Fahad University Hospital, Saudi Arabia. Cureus. 2022 Sep 23;14(9):e29489. doi: 10.7759/cureus.29489. eCollection 2022 Sep. PMID 36299951
- [Background] Al-Daghri NM, Al-Attas OS, Alokail MS, Alkharfy KM, Yousef M, Sabico SL, Chrousos GP. Diabetes mellitus type 2 and other chronic non-communicable diseases in the central region, Saudi Arabia (Riyadh cohort 2): a decade of an epidemic. BMC Med. 2011 Jun 20;9:76. doi: 10.1186/1741-7015-9-76. PMID 21689399
- [Background] Assiri AA, Alahmari KA, Alqhtani NS, AlShamrani NA, Mubarak AS, Alshehri KM, Alselmi AA. Prevalence of cardiovascular events among patients with type 2 diabetes in the west region of Saudi Arabia. Saudi Pharm J. 2022 Dec;30(12):1825-1829. doi: 10.1016/j.jsps.2022.10.012. Epub 2022 Nov 3. PMID 36601500
- [Background] Alshamiri M, Ghanaim MMA, Barter P, Chang KC, Li JJ, Matawaran BJ, Santoso A, Shaheen S, Suastika K, Thongtang N, Yusof AK. Expert opinion on the applicability of dyslipidemia guidelines in Asia and the Middle East. Int J Gen Med. 2018 Jul 18;11:313-322. doi: 10.2147/IJGM.S160555. eCollection 2018. PMID 30050317
- [Background] Cheng YJ, Imperatore G, Geiss LS, Saydah SH, Albright AL, Ali MK, Gregg EW. Trends and Disparities in Cardiovascular Mortality Among U.S. Adults With and Without Self-Reported Diabetes, 1988-2015. Diabetes Care. 2018 Nov;41(11):2306-2315. doi: 10.2337/dc18-0831. Epub 2018 Aug 21. PMID 30131397
- [Background] Yun JS, Ko SH. Current trends in epidemiology of cardiovascular disease and cardiovascular risk management in type 2 diabetes. Metabolism. 2021 Oct;123:154838. doi: 10.1016/j.metabol.2021.154838. Epub 2021 Jul 30. PMID 34333002
- [Background] Chow CK, Islam S, Bautista L, Rumboldt Z, Yusufali A, Xie C, Anand SS, Engert JC, Rangarajan S, Yusuf S. Parental history and myocardial infarction risk across the world: the INTERHEART Study. J Am Coll Cardiol. 2011 Feb 1;57(5):619-27. doi: 10.1016/j.jacc.2010.07.054. No abstract available. PMID 21272754
- [Background] Lloyd-Jones DM, Nam BH, D'Agostino RB Sr, Levy D, Murabito JM, Wang TJ, Wilson PW, O'Donnell CJ. Parental cardiovascular disease as a risk factor for cardiovascular disease in middle-aged adults: a prospective study of parents and offspring. JAMA. 2004 May 12;291(18):2204-11. doi: 10.1001/jama.291.18.2204. PMID 15138242
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- [Background] Savji N, Rockman CB, Skolnick AH, Guo Y, Adelman MA, Riles T, Berger JS. Association between advanced age and vascular disease in different arterial territories: a population database of over 3.6 million subjects. J Am Coll Cardiol. 2013 Apr 23;61(16):1736-43. doi: 10.1016/j.jacc.2013.01.054. Epub 2013 Apr 2. PMID 23500290
- [Background] Asia Pacific Cohort Studies Collaboration. Joint effects of systolic blood pressure and serum cholesterol on cardiovascular disease in the Asia Pacific region. Circulation. 2005 Nov 29;112(22):3384-90. doi: 10.1161/CIRCULATIONAHA.105.537472. Epub 2005 Nov 21. PMID 16301345
- [Background] Lowe LP, Greenland P, Ruth KJ, Dyer AR, Stamler R, Stamler J. Impact of major cardiovascular disease risk factors, particularly in combination, on 22-year mortality in women and men. Arch Intern Med. 1998 Oct 12;158(18):2007-14. doi: 10.1001/archinte.158.18.2007. PMID 9778200
- [Background] Global Cardiovascular Risk Consortium; Magnussen C, Ojeda FM, Leong DP, Alegre-Diaz J, Amouyel P, Aviles-Santa L, De Bacquer D, Ballantyne CM, Bernabe-Ortiz A, Bobak M, Brenner H, Carrillo-Larco RM, de Lemos J, Dobson A, Dorr M, Donfrancesco C, Drygas W, Dullaart RP, Engstrom G, Ferrario MM, Ferrieres J, de Gaetano G, Goldbourt U, Gonzalez C, Grassi G, Hodge AM, Hveem K, Iacoviello L, Ikram MK, Irazola V, Jobe M, Jousilahti P, Kaleebu P, Kavousi M, Kee F, Khalili D, Koenig W, Kontsevaya A, Kuulasmaa K, Lackner KJ, Leistner DM, Lind L, Linneberg A, Lorenz T, Lyngbakken MN, Malekzadeh R, Malyutina S, Mathiesen EB, Melander O, Metspalu A, Miranda JJ, Moitry M, Mugisha J, Nalini M, Nambi V, Ninomiya T, Oppermann K, d'Orsi E, Pajak A, Palmieri L, Panagiotakos D, Perianayagam A, Peters A, Poustchi H, Prentice AM, Prescott E, Riserus U, Salomaa V, Sans S, Sakata S, Schottker B, Schutte AE, Sepanlou SG, Sharma SK, Shaw JE, Simons LA, Soderberg S, Tamosiunas A, Thorand B, Tunstall-Pedoe H, Twerenbold R, Vanuzzo D, Veronesi G, Waibel J, Wannamethee SG, Watanabe M, Wild PS, Yao Y, Zeng Y, Ziegler A, Blankenberg S. Global Effect of Modifiable Risk Factors on Cardiovascular Disease and Mortality. N Engl J Med. 2023 Oct 5;389(14):1273-1285. doi: 10.1056/NEJMoa2206916. Epub 2023 Aug 26. PMID 37632466
- [Background] Vasan RS, Sullivan LM, Wilson PW, Sempos CT, Sundstrom J, Kannel WB, Levy D, D'Agostino RB. Relative importance of borderline and elevated levels of coronary heart disease risk factors. Ann Intern Med. 2005 Mar 15;142(6):393-402. doi: 10.7326/0003-4819-142-6-200503150-00005. PMID 15767617
- [Background] Joseph JJ, Deedwania P, Acharya T, Aguilar D, Bhatt DL, Chyun DA, Di Palo KE, Golden SH, Sperling LS; American Heart Association Diabetes Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Clinical Cardiology; and Council on Hypertension. Comprehensive Management of Cardiovascular Risk Factors for Adults With Type 2 Diabetes: A Scientific Statement From the American Heart Association. Circulation. 2022 Mar;145(9):e722-e759. doi: 10.1161/CIR.0000000000001040. Epub 2022 Jan 10. PMID 35000404
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Almdal T, Scharling H, Jensen JS, Vestergaard H. The independent effect of type 2 diabetes mellitus on ischemic heart disease, stroke, and death: a population-based study of 13,000 men and women with 20 years of follow-up. Arch Intern Med. 2004 Jul 12;164(13):1422-6. doi: 10.1001/archinte.164.13.1422. PMID 15249351
- [Background] Wan EYF, Yu EYT, Mak IL, Youn HM, Chan KS, Chan EWY, Wong ICK, Lam CLK. Diabetes with poor-control HbA1c is cardiovascular disease 'risk equivalent' for mortality: UK Biobank and Hong Kong population-based cohort study. BMJ Open Diabetes Res Care. 2023 Jan;11(1):e003075. doi: 10.1136/bmjdrc-2022-003075. PMID 36634978
- [Background] Laakso M, Kuusisto J. Insulin resistance and hyperglycaemia in cardiovascular disease development. Nat Rev Endocrinol. 2014 May;10(5):293-302. doi: 10.1038/nrendo.2014.29. Epub 2014 Mar 25. PMID 24663222
- [Background] Iglay K, Hannachi H, Joseph Howie P, Xu J, Li X, Engel SS, Moore LM, Rajpathak S. Prevalence and co-prevalence of comorbidities among patients with type 2 diabetes mellitus. Curr Med Res Opin. 2016 Jul;32(7):1243-52. doi: 10.1185/03007995.2016.1168291. Epub 2016 Apr 4. PMID 26986190
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Dal Canto E, Ceriello A, Ryden L, Ferrini M, Hansen TB, Schnell O, Standl E, Beulens JW. Diabetes as a cardiovascular risk factor: An overview of global trends of macro and micro vascular complications. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):25-32. doi: 10.1177/2047487319878371. Epub 2019 Nov 13. PMID 31722562
- [Background] Einarson TR, Acs A, Ludwig C, Panton UH. Prevalence of cardiovascular disease in type 2 diabetes: a systematic literature review of scientific evidence from across the world in 2007-2017. Cardiovasc Diabetol. 2018 Jun 8;17(1):83. doi: 10.1186/s12933-018-0728-6. PMID 29884191
- [Background] Ma CX, Ma XN, Guan CH, Li YD, Mauricio D, Fu SB. Cardiovascular disease in type 2 diabetes mellitus: progress toward personalized management. Cardiovasc Diabetol. 2022 May 14;21(1):74. doi: 10.1186/s12933-022-01516-6. PMID 35568946
- [Background] Alguwaihes AM, Alhozali A, Yahia MM, Abdel-Nabi T, Hassan Hatahet M, Albalkhi NI, Al Sifri S. The prevalence of cardiovascular disease in adults with type 2 diabetes mellitus in Saudi Arabia - CAPTURE study. Saudi Med J. 2023 Jan;44(1):57-66. doi: 10.15537/smj.2023.44.1.20220402. PMID 36634941
- [Background] Kalaf H, AlMesned A, Soomro T, Lasheen W, Ewid M, Al-Mohaimeed AA. Cardiovascular disease risk profile among young Saudi women of Al-Qassim, Saudi Arabia: A cross-sectional study. Int J Health Sci (Qassim). 2016 Jan;10(1):29-37. doi: 10.12816/0031214. PMID 27004055
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Alhabib KF, Batais MA, Almigbal TH, Alshamiri MQ, Altaradi H, Rangarajan S, Yusuf S. Demographic, behavioral, and cardiovascular disease risk factors in the Saudi population: results from the Prospective Urban Rural Epidemiology study (PURE-Saudi). BMC Public Health. 2020 Aug 8;20(1):1213. doi: 10.1186/s12889-020-09298-w. PMID 32770968
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Rawshani A, Rawshani A, Franzen S, Eliasson B, Svensson AM, Miftaraj M, McGuire DK, Sattar N, Rosengren A, Gudbjornsdottir S. Mortality and Cardiovascular Disease in Type 1 and Type 2 Diabetes. N Engl J Med. 2017 Apr 13;376(15):1407-1418. doi: 10.1056/NEJMoa1608664. PMID 28402770
- [Background] World health statistics 2020: monitoring health for the SDGs, sustainable development goals. Geneva: World Health Organization 2020 Licence: CC BY-NC-SA 30 IGO.
- See also: IDF Diabetes Atlas [Internet]. [cited 2024 Jul 31] — https://diabetesatlas.org/
- See also: Internet and social media users in the world 2024 | Statista [Internet]. [cited 2024 Aug 1]. — https://www.statista.com/statistics/617136/digital-population-worldwide/
- See also: Social media usage in Saudi Arabia - statistics & facts — https://www.statista.com/topics/9947/social-media-usage-in-saudi-arabia/
- See also: Prevalence of Established Cardiovascular Disease in Patients with Type 2 Diabetes Mellitus in the UK — https://link.springer.com/article/10.1007/s13300-019-00698-9
- See also: World health statistics 2021. monitoring health for the SDGs, sustainable development goals. Geneva: World Health Organization 2021. Licence: CC BY-NC-SA 30 IGO. — https://www.who.int/publications/i/item/9789240027053